CLINICAL TRIAL: NCT04556539
Title: SC10914 Monotherapy for gBRCA1/2 Mutation Advanced Ovarian Cancer Patients With at Least 2 Prior Lines of Chemotherapy: a Single Arm, Open Label, Multicenter Clinical Trial
Brief Title: Study of SC10914 in Patients With gBRCA1/2 Mutation Advanced Ovarian Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QF-SC10914-201
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2020-09

CONDITIONS: Advanced Ovarian Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SC10914 group (Experimental)
  Interventions: Drug: SC10914

INTERVENTIONS:
Drug: SC10914 — 400mg TID, oral admination on fasting condition

SUMMARY:
A phase II, multicenter, open-label, single-arm study to evaluate the efficacy, safety and pharmacokinetics of SC10914 in subjects with gBRCA1/2 mutated advanced ovarian cancer in china.

DETAILED DESCRIPTION:
A total of 104 subjects with gBRCA1/2 mutated advanced ovarian cancer is planned to be enrolled to observe the efficacy, safety and PK profile of SC10914.

The subjects oral administration SC10914 tablets 400mg on an empty stomach, three times a day, for 28 consecutive days as a treatment cycle, until disease progression (PD) or the toxicity was intolerable. PK blood samples are planned to be collected for each enrolled subject on C1D28 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent voluntarily;
2. ≥18 years old;
3. Histologically confirmed ovarian epithelial cancer, fallopian tube cancer or primary peritoneal cancer( high-grade carcinoma cancer or endometrioid carcinoma);
4. gBRCA1/2 mutation positive;
5. Had recived at least 2 prior lines of chemotherapy;
6. Platinum sensitive patients;
7. The last line of therapy befor enrollment failed；
8. ECOG≤2；

8. Had at least one measurable lesion.

Exclusion Criteria:

1. Any previous treatment with PARP inhibitor;
2. Symptomatic brain metastases;
3. Large amount of fluid in the third gap；
4. Subjects with not enough organ functional reserve at baseline, which met at least one of the following criteria： ANC<1.5×10^9/L PLT<100×10^9/L Hb<100g/L TBIL>1.5×ULN ALT, AST>2.5×ULN (without liver metastases) or ALT, AST>5×ULN (with liver metastases) Cr >1.5×ULN

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | up to 100 weeks (estimated)
  assessed by the independent imaging assessment committee (recist1.1)

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Cancer Hospital, Fujian, China